CLINICAL TRIAL: NCT02695147
Title: Direct Aortic vs Subclavian Access for TAVI: a Review of the Outcomes in the UK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Sussex County Hospital (Other)
Collaborators: National Institute for Cardiovascular Outcomes Research (Other)
Responsible Party: Principal Investigator, David Hildick-Smith, Consultant Cardiologist, Royal Sussex County Hospital
Other Study IDs: RoyalSussexTAVISCvsDA
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TAVI via Subclavian approach: Any TAVI procedure using any valve type performed via the subclavian approach
  Interventions: Procedure: TAVI
- TAVI via Direct Aortic approach: Any TAVI procedure using any valve type performed via the direct aortic approach
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI

SUMMARY:
A retrospective analysis of outcomes of all patients who received TAVI via the subclavian or direct aortic approach between January 2011 and January 2016

ELIGIBILITY:
Inclusion Criteria:

* Recieve TAVI via subclavian or direct aortic apporach in the UK

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received TAVI via the subclavian or direct aortic approach in the UK
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
MACE | Up to 5 years (average 3 years)

SECONDARY OUTCOMES:
Procedural Complications | 30 dyas post procedure

IPD SHARING:
Plan to Share IPD: No